CLINICAL TRIAL: NCT03270202
Title: The HUNT 4 PAI Study: A Randomized Controlled Intervention Study Using Wearable Devices to Promote Physical Activity
Brief Title: Wearable Devices to Promote Physical Activity
Acronym: HUNT4-PAI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: discontinuation of financial support
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016/2300
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Cardiovascular Diseases
Keywords: Exercise; Cardiorespiratory fitness; Risk factors; Monitoring, physiologic; Monitoring, ambulatory; Prognosis; Norway
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAI group (Experimental): Participants randomized to the PAI-group will receive a wearable device (Mio Slice PAI wristband) that measure heart rate continuously and via an algorithm calculates a physical activity score called PAI. The weekly goal of 100 PAI can be reached by a combination of different intensities and durations and the participants will get continuous information about their current score and amount of activity needed to reach the goal. 100 PAI is expected to approximate current guidelines of 150 minutes of moderate intensity or 75 minutes of vigorous intensity for the average participant or somewhat less if the intensity of the chosen activity is high. Proper instruction in use of the device and App will be given both oral and written after baseline testing and randomization.
  Interventions: Behavioral: PAI group; Behavioral: Usual care
- Usual care (Active Comparator): Usual care: Participants in the control group will be informed about, and encouraged to be active according to current recommendations for physical activity from the health authorities.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: PAI group — * physical activity defined as 100 weekly PAI during 1 year
  * smartphone application and a user-friendly activity wristband (Mio PAI Slice)
  Arms: PAI group
Behavioral: Usual care — Participants will be informed about, and encouraged to be active according to current recommendations for physical activity from the health authorities.

SUMMARY:
This study evaluates the effect of a new wearable device, that measures physical activity level based on heart rates, on relevant health outcomes including cardiorespiratory fitness. Half of participants will be instructed in using the Mio Slice wristband, while the other half will be requested to follow today's recommendations for physical activity.

DETAILED DESCRIPTION:
Two critical challenges precluding the full potential of physical activity in preventive healthcare are: 1) The majority of people are not sufficiently active, and 2) there is a lack of large, long-term intervention studies documenting the effect of personalized activity and improved health in the population. Using HUNT data an algorithm called Personal Activity Intelligence (PAI) has been developed. PAI was integrated in a smartphone application and user friendly wristband (Mio Slice), that measures heart rate continuously and estimates an individual threshold for total physical activity (defined as 100 weekly PAI) that is associated with reduced risk of cardiovascular disease and mortality. The primary aim of the study is to reveal whether using the wristband will increase cardiorespiratory fitness, determined by maximal oxygen uptake, after 4 months among low-fit participants. The secondary aims includes the effect on reversing cardiovascular risk factors, cardiac structure and function, adherence to physical activity and identification of barriers after 16 weeks and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participated in HUNT 3 and HUNT 4 Fitness Study
* VO2peak in HUNT4 in the lowest sex- and age-specific tertile.

Exclusion Criteria:

* Illness or disabilities that preclude completion of the study or make exercise contraindicated
* uncontrolled hypertension, arrhythmias or angina
* heart failure
* primary pulmonary hypertension
* diagnosed dementia
* chronic communicable infectious diseases
* participation in conflicting interventions

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) | 16 weeks
  Measured by ergospirometry during a maximal treadmill protocol to exhaustion

SECONDARY OUTCOMES:
Peak oxygen uptake (VO2peak) | 1 year
  Measured by ergospirometry during a maximal treadmill protocol to exhaustion
Cardiovascular risk profile (ESC Score) | 16 weeks
  Measured by blood samples and clinical data
Cardiovascular risk profile (ESC Score) | 1 year
  Measured by blood samples and clinical data
Structural and functional cardiac changes | 16 weeks
  Measured by echocardiography and CT coronary angiography
Structural and functional cardiac changes | 1 year
  Measured by echocardiography and CT coronary angiography
Quality of life | 16 weeks
  Measured by questionnaire SF-36
Quality of life | 1 year
  Measured by questionnaire SF-36
Adherence to prescribed physical activity | 16 weeks
  Measured by Mio Slice
Adherence to prescribed physical activity | 1 year
  Measured by Mio Slice
Feedback from users | 16 weeks
  Measured by interviews and feedback systems
Feedback from users | 1 year
  Measured by interviews and feedback systems

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, phd, Study Director — Norwegian University of Science and Technology; Bjarne Martens Nes, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
After the study ends all data from baseline and follow-up testing will be transferred to HUNT databank and made available for other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 6 months after study completion with no time-frame restriction.
Access Criteria: Data will be available for national and international institutions after contract with HUNT Research Center and includes a fee.